CLINICAL TRIAL: NCT07234175
Title: Comparison of a Procedural Oxygen Mask and Nasal Cannula for the Prevention of Hypoxemia During Pediatric Upper Gastrointestinal Endoscopy Under Sedation: A Single-Center Prospective Randomized Controlled Trial
Brief Title: Procedural Oxygen Mask vs Nasal Cannula in Pediatric Endoscopy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bedirhan Günel (Other Government)
Responsible Party: Sponsor-Investigator, Bedirhan Günel, Principal Investigator, Kocaeli City Hospital
Organization: Kocaeli City Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KSH-ANREA-BG-08
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Hypoxemia
MeSH Terms: conditions — Hypoxia | interventions — Cannula

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group P (Experimental): Participants will receive oxygen via a Procedural Oxygen Mask (POM) at a flow rate of 5 L/min during upper gastrointestinal endoscopy under sedation.
  Interventions: Device: Procedural Oxygen Mask
- Group N (Active Comparator): Participants will receive oxygen via a conventional nasal cannula at a flow rate of 5 L/min during upper gastrointestinal endoscopy under sedation.
  Interventions: Device: Nasal Cannula

INTERVENTIONS:
Device: Procedural Oxygen Mask — Delivers oxygen through the mouth and nose during sedation while allowing endoscope passage.
  Arms: Group P
Device: Nasal Cannula — Provides standard oxygen delivery through the nostrils during sedation.
  Arms: Group N

SUMMARY:
Upper gastrointestinal endoscopy is a commonly performed diagnostic and, when necessary, therapeutic procedure in pediatric patients for the evaluation of the esophagus, stomach, and duodenum. Additional interventions such as biopsy, foreign body removal, or polypectomy can also be performed during the same session. Sedation is generally required during the procedure, and the depth of sedation is often greater than that used for routine examinations.

Because of anatomical and physiological differences in children-such as smaller airway diameter, higher oxygen consumption, and lower functional residual capacity-the risks of upper airway obstruction, hypoxemia, and hypoventilation are higher than in adults. The passage of the endoscope through the mouth, combined with the respiratory depressant effects of sedatives and the smaller airway diameter, increases the likelihood of hypoxemia and limits the anesthesia team's access to the airway. Therefore, maintaining airway stability and optimizing oxygenation during sedation are particularly critical in pediatric patients.

Currently, several oxygen delivery methods are used during upper gastrointestinal endoscopy, including conventional nasal cannulas, high-flow nasal oxygen systems, and procedural oxygen masks. The Procedural Oxygen Mask (POM™) is a specially designed device that delivers oxygen through both the mouth and nose while allowing endoscope passage and continuous capnography monitoring. Previous studies in adults have shown that the use of POM™ or high-flow nasal oxygen reduces the incidence of hypoxemia during endoscopy. However, in children, there is a lack of randomized controlled trials directly comparing POM™ with nasal cannula use.

This single-center prospective randomized controlled trial aims to compare the effectiveness of the Procedural Oxygen Mask (POM™) and nasal cannula in preventing hypoxemia during pediatric upper gastrointestinal endoscopy under sedation. The findings are expected to contribute to safer sedation practices and improved airway management strategies in pediatric endoscopic procedures.

ELIGIBILITY:
Inclusion Criteria:

* Patients who consented to participate in the study
* Aged between 6 and 16 years
* Body weight >30 kg
* ASA physical status I-II
* Children scheduled to undergo procedural sedation for non-emergency upper gastrointestinal endoscopy

Exclusion Criteria:

* Lack of parental consent or refusal to sign the participant consent form
* History of endotracheal intubation within the past 3 months
* History of lower respiratory tract infection within the past 3 months
* History of intensive care unit (ICU) admission within the past 3 months
* Presence of a tracheostomy
* History of tracheostomy placement
* Patients with oxygen dependency due to any underlying disease
* Known pulmonary or cardiac disease
* Known congenital craniofacial anomalies
* Congenital or acquired upper airway malformations

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 114 (Estimated)
Dates: Start 2025-11-20 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Lowest SpO₂ level during procedure | From the start of sedation to end of endoscopy (typically 5-20 minutes)
  The lowest peripheral oxygen saturation (SpO₂) recorded between the initiation of sedation and the removal of the gastroscope was defined as the primary outcome.
  It was measured via continuous pulse oximetry, and when SpO₂ fluctuated, the value maintained for more than 10 seconds was recorded.

SECONDARY OUTCOMES:
Incidence of hypoxemia | During endoscopic procedure (from sedation start to endoscope removal)
  Defined as any drop in SpO₂ <94% lasting for at least 10 seconds. Based on pulse oximetry recordings.
Number of hypoxemic episodes | During endoscopic procedure
  Recurrent desaturations: counted when SpO₂ falls <94% again, at least 30 seconds after a return to ≥94%.
Duration of hypoxemia (in seconds) | During endoscopic procedure
  Time required for SpO₂ to return to ≥94% after each episode of desaturation (<94%).
Airway interventions | During endoscopic procedure
  Number of occurrences requiring airway maneuvers (chin lift, jaw thrust, or mask ventilation).
Hemodynamic complications | During endoscopic procedure
  Incidence of hypotension (>20% drop from baseline systolic BP), hypertension (>20% increase), bradycardia or tachycardia per age-specific thresholds.
Gastroenterologist satisfaction score | During endoscopic procedure
  Rated from 0 (poor sedation, interrupted) to 10 (optimal sedation).

CONTACTS AND LOCATIONS:
Overall Officials: Bedirhan Günel, MD, Principal Investigator — Kocaeli City Hospital
Locations (1):
- Kocaeli City Hospital, Kocaeli, Izmit, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Data will be made available upon reasonable request.